CLINICAL TRIAL: NCT05703607
Title: A PHASE 1/2 RANDOMIZED, OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MODIFIED RNA VACCINE AGAINST VARICELLA ZOSTER VIRUS IN HEALTHY INDIVIDUALS
Brief Title: A Study to Learn About a Modified RNA Vaccine Against Shingles in Healthy Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision made by the company
Sponsor: Pfizer (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C5031001; NCT05703607 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Shingles; Herpes Zoster Infection; Human
Keywords: Shingles; Vaccine; RNA vaccine; modRNA vaccine; Herpes zoster
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Suspensions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: SSA: Observer-blinded, Sponsor Open label SSB: Observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- SubStudy A (SSA): Group 1 (Experimental): Candidate 1, Dose Level 1, lyophilized, 0, 2 months schedule
  Interventions: Biological: Candidate 1: PF-07915234: VZV modRNA Powder for Suspension for Injection
- SSA: Group 2 (Experimental): Candidate 1, Dose Level 2, lyophilized, 0, 2 months schedule
  Interventions: Biological: Candidate 1: PF-07915234: VZV modRNA Powder for Suspension for Injection
- SSA: Group 3 (Experimental): Candidate 1, Dose Level 3, lyophilized, 0, 2 months schedule
  Interventions: Biological: Candidate 1: PF-07915234: VZV modRNA Powder for Suspension for Injection
- SSA: Group 4 (Experimental): Candidate 1, Dose Level 2, frozen, 0, 2 months schedule
  Interventions: Biological: Candidate 1: PF-07915234: VZV modRNA Suspension for Injection
- SSA: Group 5 (Experimental): Candidate 1, Dose Level 2, Frozen, 0, 6 months schedule
  Interventions: Biological: Candidate 1: PF-07915234: VZV modRNA Suspension for Injection
- SSA: Group 6 (Experimental): Candidate 2, frozen, 0, 2 months schedule
  Interventions: Biological: Candidate 2: PF-07921188: VZV modRNA Suspension for Injection
- SSA: Group 7 (Experimental): Candidate 3, Frozen, 0, 2 months schedule
  Interventions: Biological: Candidate 3: PF-07921186: VZV modRNA Suspension for Injection
- SSA: Group 8 (Active Comparator): Shingrix, 0, 2 months schedule
  Interventions: Biological: Shingrix
- SSA: Group 9 (Active Comparator): Shingrix, 0, 6 months schedule
  Interventions: Biological: Shingrix
- SSA: Group 10 (Experimental): Candidate 1, Dose level 4, lyophilized, 0, 6 months schedule (saline at month 6)
  Interventions: Biological: Candidate 1: PF-07915234: VZV modRNA Powder for Suspension for Injection
- Substudy B (SSB): Group 1 (Experimental): Candidate 2, Dose level 3, lyophilized, 0, 2 months schedule
  Interventions: Biological: Candidate 2: PF-07921188: VZV modRNA Powder for Suspension for Injection
- SSB: Group 2 (Experimental): Candidate 2, Dose level 4, lyophilized, 0, 2 months schedule
  Interventions: Biological: Candidate 2: PF-07921188: VZV modRNA Powder for Suspension for Injection
- SSB: Group 3 (Experimental): Candidate 2, Dose level 4, lyophilized, 0, 2 months schedule (saline at month 2)
  Interventions: Biological: Candidate 2: PF-07921188: VZV modRNA Powder for Suspension for Injection
- SSB: Group 4 (Active Comparator): Shingrix, 0, 2 months schedule
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Candidate 1: PF-07915234: VZV modRNA Powder for Suspension for Injection — Intramuscular injection
  Arms: SSA: Group 10; SSA: Group 2; SSA: Group 3; SubStudy A (SSA): Group 1
Biological: Candidate 1: PF-07915234: VZV modRNA Suspension for Injection — Intramuscular injection
  Arms: SSA: Group 4; SSA: Group 5
Biological: Candidate 2: PF-07921188: VZV modRNA Suspension for Injection — Intramuscular injection
  Arms: SSA: Group 6
Biological: Candidate 3: PF-07921186: VZV modRNA Suspension for Injection — Intramuscular injection
  Arms: SSA: Group 7
Biological: Shingrix — Intramuscular injection
  Arms: SSA: Group 8; SSA: Group 9; SSB: Group 4
Biological: Candidate 2: PF-07921188: VZV modRNA Powder for Suspension for Injection — Intramuscular injection
  Arms: SSB: Group 2; SSB: Group 3; Substudy B (SSB): Group 1

SUMMARY:
The purpose of this clinical study is to learn about the safety, extent of the side effects (reaction to vaccine), and immune response (your immune system's reaction) of the study vaccine called Varicella Zoster Virus modRNA (VZV modRNA). We are seeking for healthy participants 50 through 85 years of age.

This study will be conducted in 2 substudies: Substudy A (Phase 1) and Substudy B (Phase 2).

Substudy A:

This substudy is the Phase 1 portion of the study. In this substudy, participants will receive 1 of 3 VZV modRNA vaccine candidates (different construct, different dose levels and different formulation [frozen or freeze dry powder]) or the approved shingles vaccine intramuscularly.

Participants will be assigned in 1 of 10 groups in the study. Vaccination will be given either as a 2-dose series using one of two dosing schedules (either 2-months apart or 6-months apart), or (in one of the groups), as a single VZV modRNA vaccine at the first vaccination visit and saline at the second vaccination visit.

Participants will take part in this study for 8 to 12 months depending on the group they are assigned to. Some group(s) will continue into persistence-of-immunity (overtime assessment of effect of vaccine) portion of the study. Those participants assigned to these selected groups will be involved in the study for up to 5 years.

Substudy B:

This substudy is the Phase 2 portion of the study. In this part of the study, participants will receive either VZV modRNA vaccine at selected dose level/schedule/formulation or approved shingles vaccine. This selection was determined from data collected in Substudy A.

Participants will be involved in this study for up to 5 years.

ELIGIBILITY:
Substudy A: Group 1 to Group 10

Inclusion Criteria:

1. Male or female participants 50 through 69 years of age (inclusive) at the time of consent.
2. Healthy participants who are determined by clinical assessment, including medical history and clinical judgment of the investigator, to be eligible for inclusion in the study. Note: Known infection with HIV, HCV or HBV is an exclusion in Substudy A.
3. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol

Substudy A: Group 11 to Group 14

Inclusion Criteria:

1. Male or female participants 50 through 69 years of age (inclusive) at the time of consent.
2. Healthy participants who are determined by clinical assessment, including medical history and clinical judgment of the investigator, to be eligible for inclusion in the study. Note: Known infection with HIV, HCV or HBV is an exclusion in Substudy A.
3. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
5. Has a body mass index (BMI) between 18 and 35 (inclusive) kg/m2 at the screening visit.

Substudy A: Group 1 to Group 10

Exclusion Criteria:

1. History of HZ (shingles).
2. History of Guillain-Barré syndrome.
3. Known infection with HIV, HCV, or HBV.
4. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
5. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
6. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
7. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Women who are pregnant or breastfeeding.
9. Prior history of heart disease (eg, heart failure, recent coronary artery disease, cardiomyopathies, pericarditis/myocarditis).
10. Previous vaccination with any varicella or HZ vaccine.
11. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
12. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
13. Any participant who has received or plans to receive an RNA vaccine 28 days prior to Vaccination 1.
14. Participation in other interventional studies within 28 days prior to study entry or anticipated involvement through and including 6 months after the last dose of study intervention. Participation in observational studies is permitted.
15. Any screening hematology and/or blood chemistry laboratory value that meets the definition of a ≥ Grade 1 abnormality; or any abnormal bilirubin or troponin I value.
16. Screening 12-lead ECG that, as judged by the investigator, is consistent with probable or possible myocarditis/pericarditis or demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
17. Participation or planned participation in strenuous or endurance exercise within 7 days before or after each study intervention administration.
18. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

SubStudy B:

Inclusion Criteria:

1. Male or female participants 50 through 85 years of age (inclusive) at the time of consent.
2. Healthy participants who are determined by clinical assessment, including medical history and clinical judgment of the investigator, to be eligible for inclusion in the study.
3. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
5. Has a BMI between 18 and 35 (inclusive) kg/m2 at the screening visit.

Exclusion Criteria:

1. History of HZ (shingles).
2. History of Guillain-Barré syndrome.
3. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
4. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
5. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
7. Women who are pregnant or breastfeeding.
8. Prior history of heart disease (eg, heart failure, recent coronary artery disease, cardiomyopathies, pericarditis, or myocarditis).
9. Previous vaccination with any varicella or HZ vaccine.
10. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
11. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
12. Any participant who has received or plans to receive an RNA vaccine 28 days prior to Vaccination 1.
13. Participation in other interventional studies within 28 days prior to study entry or anticipated involvement through and including 6 months after the last dose of study intervention is prohibited. Participation in observational studies is permitted.
14. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
SSA: Percentage of participants reporting local reactions | For 7 days after Vaccination 1 and Vaccination 2
  Pain at the injection site, redness, and swelling as self-reported in electronic diaries.
SSA: Percentage of participants reporting systemic events | For 7 days after Vaccination 1 and Vaccination 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain, as self-reported in electronic diaries
SSA: Percentage of participants reporting adverse events | From Vaccination 1 to 4 weeks after last vaccination
  As elicited by investigational site staff
SSA: Percentage of participants reporting serious adverse events | From Vaccination 1 to 6 months after the last study vaccination
  As elicited by investigational site staff
SSA: Percentage of participants reporting medically attended adverse event | From Vaccination 1 to 6 months after the last study vaccination
  As elicited by investigational site staff
SSA: Percentage of participants with abnormal hematology and chemistry laboratory assessments | 3 days and 1 week after each vaccination
  As measured at the central laboratory
SSA: Percentage of participants with new electrocardiogram (ECG) abnormalities | 3 days and 1 week after each vaccination
  ECG abnormalities consistent with probable or possible myocarditis or pericarditis, as judged by a cardiologist
SSA: Percentage of participants with abnormal troponin I laboratory values | 3 days and 1 week after each vaccination
  as measured at the central laboratory
SSB: Percentage of participants reporting local reactions | For 7 days after Vaccination 1 and Vaccination 2
  Pain at the injection site, redness, and swelling as self-reported in electronic diaries.
SSB: Percentage of participants reporting systemic events | For 7 days after Vaccination 1 and Vaccination 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, muscle pain, and joint pain, as self-reported in electronic diaries
SSB: Percentage of participants reporting adverse events | From Vaccination 1 to 4 weeks after last vaccination
  As elicited by investigational site staff
SSB: Percentage of participants reporting serious adverse events | From Vaccination 1 to 6 months after the last study vaccination
  As elicited by investigational site staff
SSB: Percentage of participants reporting medically attended adverse events | From Vaccination 1 to 6 months after the last study vaccination
  As elicited by investigational site staff

SECONDARY OUTCOMES:
SSA: Geometric mean concentrations (GMCs) of glycoprotein E antibodies in proportion of evaluable immunogenicity participant | At baseline (before vaccination 1), at 1- and 4-weeks after each vaccination and 6-months after last vaccination
  As measured at the central laboratory
SSA: Geometric mean fold rise (GMFR) from before vaccination to each subsequent timepoint in evaluable immunogenicity participants | At baseline (before vaccination 1), at 1- and 4-weeks after each vaccination and 6-months after last vaccination
  As measured at the central laboratory
SSA: Proportion of evaluable immunogenicity participants with vaccine response in glycoprotein E antibodies from baseline to each subsequent timepoint | At baseline (before vaccination 1), at 1- and 4-weeks after each vaccination and 6-months after last vaccination
  As measured at the central laboratory
SSB: Geometric mean concentrations (GMCs) of glycoprotein E antibodies in proportion of evaluable immunogenicity participant | At baseline (before vaccination 1), at 4-weeks after each vaccination and 6-months after last vaccination
  As measured at the central laboratory
SSB: Geometric mean fold rise (GMFR) from before vaccination to each subsequent timepoint in evaluable immunogenicity participants | At baseline (before vaccination 1), at 4-weeks after each vaccination and 6-months after last vaccination
  As measured at the central laboratory
SSB: Proportion of evaluable immunogenicity participants with vaccine response in glycoprotein E antibodies from baseline to each subsequent timepoint | At baseline (before vaccination 1), at 4-weeks after each vaccination and 6-months after last vaccination
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (35):
  - Tri-City Cardiology, Gilbert, Arizona
  - Aventiv Research Inc., Mesa, Arizona
  - Stanford University Medical Center, Palo Alto, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - GW Vaccine Research Unit, Washington D.C., District of Columbia
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - West Valley Cardiology Services, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - University of Iowa, Iowa City, Iowa
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Centennial Medical Group, Columbia, Maryland
  - Associates in Cardiology, PA, Silver Spring, Maryland
  - C.S. Mott Clinical Research Center (CRC), Detroit, Michigan
  - Henry Ford St. John Hospital, Grosse Pointe Woods, Michigan
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - University of Nevada School of Medicine - Reno, Reno, Nevada
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - Tisch Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Wilmington Health, PLLC (Cardiologist), Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Columbus Cardiovascular Associates, Inc., Columbus, Ohio
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5031001